CLINICAL TRIAL: NCT06037044
Title: The Effect of Sensory Integration Balance Training Compared With Traditional Balance Training for Children With Acquired Brain Injury (ABI)
Brief Title: The Effect of Sensory Integration Balance Training on Children With ABI
Acronym: ABI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Afrah Almuwais, Assistant prof, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB log #22-0364
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Children With Acquired Brain Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor will be blinded to group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory integration therapy for balance and gait (Experimental): Sensory integration walking pathway with obstacles x 10 and standing on one leg with eyes open and eyes closed 5-10 sec
  Interventions: Other: Sensory integration therapy for balance and gait training; Other: Traditional Physiotherapy for balance and gait training
- Traditional Physiotherapy for balance and gait (Active Comparator): Walking pathway with obstacles x 10 and standing on one leg with eyes open 5-10 sec
  Interventions: Other: Sensory integration therapy for balance and gait training; Other: Traditional Physiotherapy for balance and gait training

INTERVENTIONS:
Other: Sensory integration therapy for balance and gait training — Sensory integartion Walking pathway with obstacles x10 rep, standing on one leg with eyes op5-10 sec x10 rep)
Other: Traditional Physiotherapy for balance and gait training — Traditional Physiotherapy walking pathway with obstacles x10 rep, standing on one leg with eyes open 5-10 sec x10 rep

SUMMARY:
This study aim to investagte the effectivness of sensory integartion balance training during gait training with obstecles and stimulation to different sensation, in comparission to gait training with obstecles without sensory stimulation among children with acuired brain injury

ELIGIBILITY:
Inclusion Criteria:

* Children with ABI, able to walk with or without assistance, GMFCS level I-III, aged 4-12 years old, with subjective symptoms of balance impairments, fear of falling and/or history of falls

Exclusion Criteria:

* Botox injections or tendon release surgery in the past six months

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Pediatric balance scale (PBS) | One week before and after training then one month after training
  It was developed as a balance measure for children. The PBS measure can be performed without specialized equipment and is quickly and easily administered. The PBS has been used to measure the functional balance skills for school-age children with mild-to-moderate motor impairments. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points. These items include moving from a seated to a standing position, moving from a standing position to a sitting position, transfer, standing without support, sitting without support, standing with eyes closed, standing with feet together, standing with one foot in front of the other, standing on one foot, rotating 360 degrees, turning to look back, picking up an object off the floor, placing alternate foot on step or footrest, and reaching forward with an extended arm.
Gross motor functional measure (GMFM) | One week before and after training then one month after training
  It is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. It has 88 items to explore motor ability in five dimensions; lying and rolling, sitting, crawling and kneeling, standing, and walking, running and jumping
Timed up and go (TUG) | One week before and after training then one month after training
  It is a simple evaluative test used to measure functional mobility and show how safely a patient can move around. The test requires a subject to stand up, walk 3 m (10 ft), turn, walk back, and sit down while timing.
Obstacle Test | One week before and after training then one month after training
  It is a timed walking test. Time is calculated while the child is walking stepping over two obstacles and walking around a basket. The pathway is 8.5 meter and the start and end lines are marked. Time is calculating as the child walking between the lines and accomplishing the obstacles. Hight of the obstacle is 15% of the child leg length, while the width is 10%. The basket was around 56 centimeters in width and 69.5 centimeters in length. The child should stand behind the start line and walk in a straight line then step over the obstacles, walk around one side of the basket then pass the end line.

SECONDARY OUTCOMES:
The Pediatric Quality of Life Inventory (PedsQL) | one week before and after training then one month after training
  It is a brief measure of health-related quality of life in children and young people. The measure is either Proxy Report or Self-Report. It has 23 items comprise four Generic Core Scales: physical functioning, emotional functioning, social functioning, school functioning.
One min sit to stand test (1-MSTST) | one week before and after training then one month after training
  The 1-MSTST typically involves an armless chair and the performance of as many sit-to-stand actions as possible in 1 min without using the upper limbs

CONTACTS AND LOCATIONS:
Locations (1):
- King abdullah bin abdulaziz university hospital, Riyadh, Saudi Arabia